CLINICAL TRIAL: NCT06120582
Title: An Open-label, Non-comparative, Single Dose-Escalation Study of the Safety, Pharmacodynamics and Efficacy of ANB-002 in Patients With Hemophilia B
Brief Title: Study of the Safety, Pharmacodynamics and Efficacy of ANB-002 in Patients With Hemophilia B (SAFRAN)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANB-002-1
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive ANB-002 (arvenacogene sanparvovec) at a dose 1. Follow-up for the assessment of dose-limiting toxicity (DLT) will be carried out for 28 days. If no DLT events are observed in the subject of Cohort 1, the following subjects will be included in Cohort 1.
  Interventions: Genetic: ANB-002, dose 1
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive ANB-002 (arvenacogene sanparvovec) at a dose 2. The decision to continue enrolling in Cohort 1 or dosing in Cohort 2 will be made at the IDMC meeting. After the IDMC makes a decision regarding the dosing in Cohort 2 subjects, the next subject will be included in Cohort 2. If no DLT events are observed in the subject of Cohort 2, the following subjects will be included in Cohort 2.
  Interventions: Genetic: ANB-002, dose 2
- Cohort 3 (Experimental): Subjects in Cohort 3 will receive ANB-002 (arvenacogene sanparvovec) at a dose 3. The decision to continue enrolling in Cohort 2 or dosing in Cohort 3 will be made at the IDMC meeting.
  Interventions: Genetic: ANB-002, dose 3
- Cohort 4 (Experimental): Exploratory cohort. Subjects in Cohort 4 (with anti-AAV5 antibodies and/or hepatitis B in anamnesis) will receive ANB-002 (arvenacogene sanparvovec) at the dose 3.
  Interventions: Genetic: ANB-002, dose 3

INTERVENTIONS:
Genetic: ANB-002, dose 1 — Adeno-associated viral vector carrying the FIX gene single infusion at dose 1.
  Other Names: arvenacogene sanparvovec
  Arms: Cohort 1
Genetic: ANB-002, dose 2 — Adeno-associated viral vector carrying the FIX gene single infusion at dose 2.
  Other Names: arvenacogene sanparvovec
  Arms: Cohort 2
Genetic: ANB-002, dose 3 — Adeno-associated viral vector carrying the FIX gene single infusion at dose 3.
  Other Names: arvenacogene sanparvovec
  Arms: Cohort 3; Cohort 4

SUMMARY:
The goal of this multicenter, two-stage, open-label study is to investigate the safety, immunogenicity, and efficacy of ANB-002 in subjects with hemophilia В. The study will have a dose-escalation design with elements of phase I/II seamless adaptive design.

DETAILED DESCRIPTION:
The study design includes ANB-002 dose escalation in at three cohorts. In Cohort 1, the subject is treated with a single dose of ANB-002 (dose 1) administered as an intravenous infusion. Follow-up for the assessment of dose-limiting toxicity (DLT) will be carried out for 28 days. If no DLT events are observed in the subject of Cohort 1, the following subjects will be included in Cohort 1.

In Cohort 2, the subjects are treated with a single dose of ANB-002 (dose 2). In Cohort 3, the subject are treated with a single dose of ANB-002 (dose 3).

The decision to continue enrolling in cohorts will be made at the Independent Data Monitoring Committee (IDMC) meeting. After the IDMC makes a decision regarding the dosing subjects, further enrolment to the cohort will be carried out.

Based on the data from the follow-up period of subjects included in Сohorts 1-3, a potential therapeutic dose for further study will be determined and additional patients will be included to recieve this dose.

In exploratory Cohort 4 patients with anti-AAV5 antibodies and/or hepatitis B in anamnesis will be included. These subjects will recieve the dose 3 of ANB-002.

The total duration of participation of one subjects in the study will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male with hemophilia B.
2. Age ≥18 years.
3. FIX activity at screening ≤2% without FIX inhibitor.
4. ≥150 previous exposure days of treatment with FIX concentrates.

Exclusion Criteria:

1. Previous gene therapy.
2. Other blood or hematopoietic disorders.
3. Positive Anti-AAV5 antibodies (for Cohorts 1-3).
4. Diagnosed HIV-infection, not controlled with anti-viral therapy.
5. Hepatitis B (for Cohorts 1-3), acute or chronic hepatitis C.
6. Any active systemic infections or recurrent infections requiring systemic therapy at screening.
7. Any other disorders associated with severe immunodeficiency.
8. Significant hepatic disorders (liver cirrhosis, liver fibrosis, etc).
9. Malignancies with remission <5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in FIX activity from baseline | 12 months; final assessment - 5 years
Proportion of subjects with adverse reactions | 12 months; final assessment - 5 years

SECONDARY OUTCOMES:
Changes in FIX activity | 5 years
Annualized use of FIX concentrates | 5 years
Annualized bleeding rate | 5 years
Annualized rate of bleedings requiring therapy with FIX concentrates | 5 years
Changes in Haemo-A-QoL (Hemophilia-Specific Quality of Life) scores from baseline | 5 years
  Haemo-A-QoL is a quality of life (QoL) assessment instrument for patients with haemophilia, including the domains of consequences of bleeding, emotional impact, physical functioning, role functioning, treatment concern, and worry. Using scale overall score ranges from 0 to 100.The high score represent low quality of life.
Changes in EuroQol-5D-3L (European Quality of Life Questionnaire) scores from baseline | 5 years
  The EQ-5D-5L descriptive system of health-related QoL states consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ-5D-5L VAS overall score ranges from 0 to 100. A higher score is considered to be more favorable.
Changes in SF-36 (Short Form-36) scores from baseline | 5 years
  SF-36 is a questionnaire for evaluating health-related QoL (Quality of Life). The 36 questions are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. SF-3 overall score ranges from 0 to 100. The lower the score the more disability.
Response duration based on FIX activity | 5 years
Evaluation of the condition of joints based on the Hemophilia Joint Health Score (HJHS) | 5 years
  Hemophilia Joint Health Score (HJHS) is the assessment system of joints in patients with haemophilia. Each joint (knee, elbow and ankle) receives a numeric score, which can be compared to itself over time to determine whether a joint is showing degeneration. The maximum score for an individual index joint is 20. Gait is scored 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, MD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (17):
- Belarus (2):
  - Republican Scientific and Practical Center for Radiation Medicine and Human Ecology, Homyel
  - Minsk Scientific and Practical Center for Surgery, Transplantology and Hematology, Minsk
- Russia (15):
  - State Autonomous Institution for Healthcare "Chelyabinsk Regional Clinical Hospital", Chelyabinsk
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Gatchina
  - Kuzbass Clinical Hospital named after S.V. Belyaev, Kemerovo
  - Federal State Budgetary Organization of Science "Kirov Research Institute of Hematology and Blood Transfusions of Federal Medical Biological agency", Kirov
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Clinical Diagnostics for Hematology and Hemostasis Disorders), Moscow
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Traumatology and Reconstructive and Restorative Orthopedics for Patients with Hemophilia), Moscow
  - Federal Budgetary Institution "Moscow City Clinical Hospital named after S. P. Botkin", Moscow
  - LLC "Medis", Nizhny Novgorod
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Russian Research Institute of Hematology and Transfusiology Federal State Institution of Federal Medical and Biological Agency, Saint Petersburg
  - City Polyclinic №37, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Healthcare of the Russian Federation, Samara
  - State Institution "Komi Republican Oncological Dispensary", Syktyvkar
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Healthcare of the Russian Federation, Ufa

REFERENCES:
- See also: Related Info — https://library.ehaweb.org/eha/2025/eha2025-congress/4161329/nadezhda.zozulya.arvenacogene.sanparvovec.a.novel.option.for.hemophilia.b.gene.html?f=menu%3D6%2Abrowseby%3D8%2Asortby%3D2%2Amedia%3D3%2Ace_id%3D2882%2Aot_id%3D31584%2Amarker%3D5844%2Afeatured%3D19595